CLINICAL TRIAL: NCT01242670
Title: A Phase 3 Study to Assess the Immunogenicity, Safety, and Consistency of Lot Manufacture of Ross River Virus (RRV) Vaccine in Healthy Male and Female Subjects 16 Years of Age and Older
Brief Title: Ross River Virus (RRV) Vaccine Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 880801
Record Dates: First submitted 2010-11-15; First posted 2010-11-17 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2013-01

CONDITIONS: Prophylaxis of Ross River Virus Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ross River Virus Vaccine (Experimental): Subjects will be randomized in equal numbers (1:1:1) to receive one of three different lots of the vaccine on Day 1, Day 22 and Day 181. (The study is blinded with regard to which vaccine lot is administered to a subject but all subjects will receive 3 injections with a 2.5 µg aluminum hydroxide adjuvanted dose of RRV vaccine.)
  Interventions: Biological: Ross River Virus Vaccine

INTERVENTIONS:
Biological: Ross River Virus Vaccine — Ross River Virus Vaccine (Formalin Treated, UV Inactivated, Vero Cell-Derived) with Aluminum Hydroxide Adjuvant

SUMMARY:
The purpose of the study is to verify the safety and adequacy of the immune response produced by a 2.5 µg, adjuvanted (aluminium hydroxide) dose of Ross River Virus (RRV) vaccine and to demonstrate the consistency of manufacture of 3 separate lots of RRV vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 16 to 59 years of age on the day of screening (for Stratum A only)
* Subject is 60 years of age or older on the day of screening (for Stratum B only)
* Subject and, if applicable, subject's parent(s)/legal guardian(s) has (/have) an understanding of the study and its procedures, agree to its provisions, and give written informed consent prior to study entry
* Subject provides written assent according to his/her age, if applicable
* Subject is generally healthy as determined by the investigator's clinical judgment based upon medical history and physical examination
* Subject is physically and mentally capable of participating in the study and following study procedures
* Subject agrees to keep a daily record of symptoms for the duration of the study
* If female of childbearing potential - subject has a negative urine pregnancy test result within 24 hours of the scheduled first vaccination and agree to employ adequate birth control measures for the duration of the study

Exclusion Criteria:

* Subject has a Body Mass Index > 35.0
* Subject has an elevated blood pressure at screening of > 159 mmHg systolic and/or > 99 mmHg diastolic while seated and at rest and confirmed by 2 additional measurements taken at least 30 minutes apart (while seated and at rest)
* Subject has any inherited or acquired immune deficiency
* Subject has or has a recent history of significant neurological, cardiovascular, respiratory (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder
* Subject has a history of arthritis (including RRV disease, joint swelling, tenderness, warmth or erythema) on more than one occasion, not related to trauma (including running) or any episode of non-trauma related arthritis within the previous 6 months
* Subject has a disease or is currently undergoing a form of treatment or was undergoing a form of treatment within 30 days prior to study entry that could be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (> 800 μg/day of beclomethasone dipropionate or equivalent), corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs
* Subjects has received any vaccination within 30 days prior to study entry
* Subject has received a blood transfusion or immunoglobulins within 90 days prior to study entry
* Subject has donated blood or plasma within 30 days prior to study entry
* Subject has a history of any vaccine related contraindicating event (eg, anaphylaxis, allergy to components of the test vaccine, other known contraindications)
* Subject has a dermatologic condition or tattoos which may interfere with injection site reaction rating
* Subject has participated in another clinical study involving an investigational drug, biological product or device within 30 days prior to enrollment in this study or is scheduled to participate in another clinical study involving an investigational drug, biological or device during the course of this study
* Subject has functional or surgical asplenia
* Subject has a known or suspected problem with alcohol or drug abuse
* Subject is a member of the team conducting this study or is in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees of the investigator or site personnel conducting this study
* Subject is pregnant or lactating

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1968 (Actual)
Dates: Start 2011-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Immune response measured by Ross River Vaccine (RRV)-specific neutralizing titer 21 days after the 3rd vaccination as determined by RRV microneutralization (μNT) assay | 21 days after 3rd vaccination
Rate of subjects with a RRV-specific neutralizing titer | 21 days after 3rd vaccination
  Rate of subjects with a RRV-specific neutralizing titer 21 days after the third vaccination as determined by RRV microneutralization (μNT) assay
Frequency and severity of injection site and systemic reactions within 7 days of any study vaccination | Within 7 days of any study vaccination

SECONDARY OUTCOMES:
Rate of subjects with a RRV-specific neutralizing titer | 21 days after 1st + 2nd vaccination and 180 days after 1st + 3rd vaccination
Rate of subjects with seroconversion | 21 days after 1st, 2nd + 3rd vaccination and 180 days after 1st + 3rd vaccination
  Seroconversion is defined as a positive RRV-specific neutralizing titer after vaccination (>= 1:10) when RRV-specific neutralizing titer at baseline is < 1.4 or a minimum 4-fold RRV-specific neutralizing titer increase as compared to baseline
Immune response measured by RRV-specific neutralizing titer | 21 days after 1st + 2nd and 180 days after 1st + 3rd vaccination
Fold increase of RRV-specific neutralizing titer | 21 days after 1st, 2nd + 3rd vaccination and 180 days after 1st + 3rd vaccination
  Fold increase as compared to baseline
Rate of subjects with a RRV-specific immunoglobulin G (IgG) titer | 21 days after 1st, 2nd + 3rd vaccination and 180 days after 1st + 3rd vaccination
Rate of subjects with seroconversion (defined as a positive RRV-specific IgG) titer after vaccination | 21 days after 1st, 2nd + 3rd vaccination and 180 days after 1st + 3rd vaccination
Immune response measured by RRV-specific IgG titer | 21 days after 1st, 2nd + 3rd vaccination and 180 days after 1st + 3rd vaccination
Fold increase of RRV-specific IgG titer | 21 days after 1st, 2nd + 3rd vaccination and 180 days after 1st + 3rd vaccination
  Fold increase as compared to baseline
Frequency and severity of any systemic reactions | Within first 21 days of study vaccination
Frequency and severity of any injection site reactions | Within first 21 days following a study vaccination
Frequency and severity of any adverse event | During entire study period
Rate of subjects experiencing arthritis associated with one or more of the systemic symptoms consistent with RRV disease | Occurring at least 3 days after vaccination and lasting for more than 3 weeks
  Arthritis is defined as soft tissue "synovitic"swelling, ie joint effusion or synovial tissue thickening, or both, with or without pain localized to the affected joint.
  Symptoms consistent with RRV disease include fever, fatigue, malaise, rash, arthralgia, myalgia, lymphadenopathy, splenomegaly, sore throat, diarrhea, paresthesia, headache, neck stiffness, and photophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Geisberger, MD, Study Director — Baxter Innovations GmbH
Locations (17):
- Australia (17):
  - Holdsworth House, Byron Bay, New South Wales
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - St. Vincents Hospital, Darlinghurst, New South Wales
  - National Centre for Immunisation Research & Surveillance, The Children´s Hospital Westmead, Westmead, New South Wales
  - AusTrials Pty Limited, Auchenflower, Queensland
  - Wesley Research Institute Clinical Trials Centre, Auchenflower, Queensland
  - AusTrials Pty Limited, Caboolture, Queensland
  - James Cook University, Cairns, Queensland
  - Q-Pharm Pty Limited, Herston, Queensland
  - QPID Clinical Trials Centre, Royal Children´s Hospital, Herston, Queensland
  - Dept of Microbiology & Infectious Diseases, Bedford Park, South Australia
  - Melbourne Street, North Adelaide, South Australia
  - Barwon Health - The Geelong Hospital, Dept Clinical & Biomedical Sciences, Geelong, Victoria
  - Centre for Clinical Studies, Heidelberg, Victoria
  - Emeritus Research, Malvern East, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia

REFERENCES:
- [Derived] Wressnigg N, van der Velden MV, Portsmouth D, Draxler W, O'Rourke M, Richmond P, Hall S, McBride WJ, Redfern A, Aaskov J, Barrett PN, Aichinger G. An inactivated Ross River virus vaccine is well tolerated and immunogenic in an adult population in a randomized phase 3 trial. Clin Vaccine Immunol. 2015 Mar;22(3):267-73. doi: 10.1128/CVI.00546-14. Epub 2014 Dec 24. PMID 25540268